CLINICAL TRIAL: NCT03085147
Title: A Phase I/II Study of the Fluorescent PARP1 Binding Imaging Agent PARPi-FL in Patients With Oral Squamous Cell Carcinomas
Brief Title: A Dye for the Detection of Cancer of the Tongue and Mouth
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 15-336
Record Dates: First submitted 2017-03-15; First posted 2017-03-21 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Oral Squamous Cell Carcinoma (OSCC)
Keywords: Tongue; Mouth; Fluorescent PARP1 Binding Imaging Agent; PARPi-FL; 15-336
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — olaparib

STUDY DESIGN:
Intervention Model Description: This is an open label, investigator initiated single arm phase I/II study. The concentration for imaging OSCC is defined in Phase I. Phase II will then use this concentration to obtain preliminary data on the sensivity of PARPi-FL to detect and delinate OSCC.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Fluorescent PARPi Binding Imaging Agent PARPi-FL (Experimental): In the phase I of the study, increasing concentrations of PARPi-FL will be used in up to 12 patients with OSCC to determine concentration that results in the highest contrast between tumor and normal mucosa. Dose escalation will be performed in groups of three patients until image contrast decreases, side effects are noted or the concentration of PARPi-FL exceeds 1μM. Imaging will be performed in the Department of Surgery during a presurgical visit including clinical examination of the oral cavity. In the phase II part of the study the concentration of PARPi-FL determined in phase I will be used to image 18 patients with OSCC on the day of surgery. Imaging findings will be correlated with histopathologic findings in the surgically resected specimens.
  Interventions: Drug: Olaparib

INTERVENTIONS:
Drug: Olaparib — For PARRi-FL, imaging patients will first gargle a solution of PARRi-FL for 1 min, then spit out this solution and gargle with a cleaning solution (the solvent used for PARRi-FL) for 1 min. Then fluorescence imaging of the oral cavity and pharynx will be performed with an endoscope. The intensity and extent of the fluorescence signal will be recorded by one of the investigators for the tumor and adjacent normal mucosa.
  Other Names: PARPi

SUMMARY:
The purpose of this study is to test if an investigational dye, called PARPi-FL, can be used to detect this type of cancer. This will be the first time that PARPi-FL is being tried in people. First, the investigators will test the safety of PARPi-FL at different doses to find out what effects, if any, it has on people. The investigators will also see which amount of PARPi-FL is best suited to detect cancers of the mouth and tongue.

ELIGIBILITY:
Inclusion Criteria:

* Patient is ≥ 18 years old
* Histologically or cytologically proven squamous cell carcinoma of the oral cavity or pharynx (OSCC)
* Scheduled to undergo surgery at MSK
* Any tumor stage, any N, M0
* ECOG performance status 0 or 1

Exclusion Criteria:

* Any surgical therapy in the area of the oral cavity or pharynx within the last 2 weeks
* Prior or ongoing treatment with a PARP1 inhibitor
* Known hypersensitivity to Olaparib
* Known hypersensitivity to PEG Eligibility criteria will be assessed by an experienced oral surgeon, typically the Co-PI of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2017-03-15 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
escalating levels of toxicity (CTCAE v 4.0) | 1 year
  toxicity data relevant to study interventions (CTCAE v 4.0)

CONTACTS AND LOCATIONS:
Overall Officials: Heiko Schoder, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge (Consent Only), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Consent only), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Consent only), Montvale, New Jersey
  - Memorial Sloan Kettering Suffolk-Commack (Consent only), Commack, New York
  - Memorial Sloan Kettering Westchester (Consent Only), Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau (Consent only), Rockville Centre, New York

REFERENCES:
- [Derived] Demetrio de Souza Franca P, Kossatz S, Brand C, Karassawa Zanoni D, Roberts S, Guru N, Adilbay D, Mauguen A, Valero Mayor C, Weber WA, Schoder H, Ghossein RA, Ganly I, Patel SG, Reiner T. A phase I study of a PARP1-targeted topical fluorophore for the detection of oral cancer. Eur J Nucl Med Mol Imaging. 2021 Oct;48(11):3618-3630. doi: 10.1007/s00259-021-05372-6. Epub 2021 May 5. PMID 33954826
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm